CLINICAL TRIAL: NCT06017713
Title: Direct Transcranial Stimulation With Direct Current Associated With Symptom Provocation in the Management of Patients With Resistant Obsessive Compulsive
Brief Title: tDCS Associated With Symptom Provocation in the Management of Patients With Resistant Obsessive Compulsive Disorder
Acronym: PPSTDCS-TOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01148-37
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tDCS + symptoms provocation (Experimental)
  Interventions: Behavioral: tDCS + symptoms provocation

INTERVENTIONS:
Behavioral: tDCS + symptoms provocation — The treatment consists of 10 sessions of tDCS. Each tDCS session lasts 30 minutes at an intensity of 2mA and is preceded by a provocation of symptoms.

SUMMARY:
This is a single-center study about patients with severe resistant OCD.

Main assumption is that performing 10 tDCS sessions with the anode positioned at the level of the right orbitofrontal cortex, and the cathode at the level of the supplementary motor area, associated with the provocation of symptoms before each session is effective in the reduction in obsessive-compulsive symptoms.

After the inclusion visit, the treatment period is provided from D1 to D12 (one session per day from Monday to Friday, for two consecutive weeks, i.e. a total of ten sessions). Each tDCS session lasts 30 minutes at an intensity of 2 mA and is preceded by symptom provocation using a standardized procedure performed by trained personnel.

The patients are then assessed on D42 and D102 (i.e. 1 month and 3 months after the end of the tDCS sessions).

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from OCD evolving for at least 2 years diagnosed according to DSM-V criteria;
* Patient with good insight, defined by a score less than or equal to 18 at the threshold of delusions on the BABS (Brown Assessment of Beliefs Scale) insight scale;
* Absence of a current depressive episode (MADRS score < 21) or suicidal risk (MADRS score item 10 < 3);
* Absence of epileptic pathology;
* Chronic obsessive-compulsive disorder defined by a total YBOCS score > 20, or a subscale score > 15;
* Drug-resistant obsessive-compulsive disorder despite treatment with:

  1. at least 2 antidepressants of the IRS type at an effective dose and for a sufficient duration
  2. and/or Behavioral and Cognitive therapy for at least 1 year;
* Therapeutic stability (antidepressants) for more than 12 weeks without significant improvement. This treatment, at a fixed dose, will be maintained during the study;
* Patient aged between 18 and 70 included
* Patient who has given his/her informed consent after having received written information on the planned procedure;
* Patient benefiting from social security or by benefiting through a third party.

Exclusion Criteria:

* Woman of childbearing age without effective means of contraception (hormonal/mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total oophorectomy)
* Pregnant or nursing woman;
* Patient hospitalized under duress (SPDT, SPDRE);
* Patient under guardianship or curatorship;
* Patient with another DSM-V Axis 1 diagnosis (Schizophrenic Disorder, Bipolar Disorder, Substance Abuse or Substance Dependence).

Generalized anxiety disorder, social phobia, nicotine addiction and history of major depressive episodes are not exclusion criteria. Axis I comorbidity will be explored using MINI 5.0.0. ;

* Patient suffering from a current depressive episode;
* Patient at risk of suicide;
* Patient with skin lesions on the scalp;
* History of head trauma;
* Patient with an intracerebral metal object
* Patient with a pacemaker;
* Presence of epileptic pathology;
* Patient in an emergency situation or unable to give personal consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
YBOCS scale | 3,5 months
  The primary endpoint corresponds to the change in the score on the YBOCS scale between the inclusion visit (Day 0) and the Day 42 visit.
  A score of 0 corresponds to the absence of OCD and a score of 40 to maximum severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France